CLINICAL TRIAL: NCT00506064
Title: Melatonin Postoperative Sleep Study in Breast Cancer Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated due to low accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DM02-563
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Results first posted 2011-01-25 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Sleep; Melatonin; Placebo; Survey; Postoperative Srejic Sleep SAT Survey
MeSH Terms: conditions — Breast Neoplasms | interventions — Melatonin; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Melatonin (Experimental): 0.15 mg/kg capsules by mouth daily
  Interventions: Drug: Melatonin; Behavioral: Questionnaire
- Placebo (Placebo Comparator): Starch capsules by mouth daily
  Interventions: Drug: Placebo; Behavioral: Questionnaire

INTERVENTIONS:
Drug: Melatonin — 0.15 mg/kg by mouth (PO) Daily
  Arms: Melatonin
Drug: Placebo — Two, three, or four starch tablet or capsules before bed
  Arms: Placebo
Behavioral: Questionnaire — Sleep study surveys, two per day completed each evening, lasting 10 minutes
  Other Names: Survey; Insomnia Syndrome Questionnaire; Postoperative Srejic Sleep SAT Survey Questionnaire

SUMMARY:
Primary Objective:

To evaluate the impact of postoperative exogenous nocturnal melatonin supplementation on the early regulation of the sleep-wake cycle and its clinical impact (subjective improvement of the quality of sleep and reduction of cardiopulmonary events) during the first postoperative week following anesthesia and surgery in older breast cancer patients receiving a unilateral segmental mastectomy with or without intraoperative lymph node mapping, sentinel node biopsy and axillary node dissection.

Secondary Objective:

To collect data and validate the Postoperative Srejic Sleep SAT Survey Questionnaire (SAT implies relative subjective satisfaction of the patient's sleep in a scaled score out of 100 with 100 being the highest degree of satisfaction).

DETAILED DESCRIPTION:
Melatonin is produced by a small gland in the brain called the pineal gland. During times of stress, use of certain medications, and increasing age, melatonin production may be disrupted or weakened. This may cause sleep disturbance. Many of the drugs used for pain, anesthesia, or cancer treatment may affect the body's natural secretion of melatonin.

Participants in this study will be randomly assigned (as in the toss of a coin) to one of two treatment groups. Participants in one group will receive melatonin. Participants in the other group will receive a placebo. A placebo is a substance that looks like the study drug, but which has no active ingredients. There is an equal chance of being in either group. Neither you nor the study doctor will know to which group you are assigned. You will take either two, three, or four capsules 30 minutes before you go to bed. You will go to bed at about the same time each day (around 10:00PM). The number of capsules will be prescribed according to your body weight.

Researchers will attach two monitors to you while you are sleeping to test for changes during sleep. An actigraph wrist monitor will be worn on the non-dominant wrist (to measure sleep movement and patterns). A pulse oximeter will be worn on the opposite hand/finger (to measure the amount of oxygen in the blood). You may use these devices as an inpatient or outpatient at home.

Each day of the study (for one week after the operation and anesthesia) you will fill out 1-2 questionnaires depending on the day. The researchers will ask questions about your last night's sleep and how you are feeling. The questionnaires will be filled out each evening. This will take less than 10 minutes.

If on Day 4 you require any additional sleep medicine or have been experiencing any unpleasant side effects of melatonin, you may remove yourself from the study. The entire length of this study is made up of the one week after your surgery. Should you take any other sleep aids during the time of the study, please tell the research staff as your questionnaire data cannot then be used for this study.

You will visit your cancer doctor and the study doctor at least one time after your surgery. This follow-up visit will be coordinated with your surgical postoperative visit. Researchers may go over some parts of the questionnaires and retrieve the actigraph and pulse oximeter from you.

This is an investigational study. Melatonin has not gone through the FDA approval process. However, melatonin supplements are commercially available in over-the-counter form. Forty patients will take part in this study. All will be enrolled at UTMDACC.

ELIGIBILITY:
Inclusion Criteria:

1. Breast cancer patients having a unilateral segmental mastectomy, with or without intraoperative lymph node mapping, sentinel node biopsy, and axillary node dissection
2. Ages >= 40 years
3. American Society of Anesthesiology (ASA) physical status classification of preoperative functioning) 1-4 levels are acceptable
4. Willing and able to give written informed consent
5. Willing and able to complete questionnaires
6. Not currently taking benzodiazepine medication for insomnia.

Exclusion Criteria:

1. Autoimmune diseases: rheumatoid arthritis, systemic lupus, or other collagen vascular disease
2. Alcoholics
3. Seizure disorder
4. Thyroid disease
5. Pregnant or lactating patients (effects not known in pregnancy)
6. Renal/hepatic failure (if ood urea nitrogen (BUN) or creatinine (Cr) >2.5* Upper limit of normal (ULN); Bili or aspartate aminotransferase (AST) or alanine aminotransferase (ALT)>2.5* ULN)
7. Dementia/poor compliance
8. Manic/psychotic patients
9. Children/adults under 40 yrs
10. Movement disorders (ex. restless leg syndrome)
11. Tremor disorder (ex. parkinsonism)
12. Chronic benzodiazepine use for sleep (>4 times per week )
13. Designated preop medications including melatonin for sleep

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2004-02; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Una Srejic, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 01/26/07 through 10/10/07. All participants recruited at UT MD Anderson Cancer Center.
Pre-assignment Details: Protocol terminated early as unable to accrue cases. There were four patients accrued of which three were not assigned, therefore data available for only one case.
Period: Overall Study
Arm/Group | Melatonin | Placebo
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Melatonin | Placebo | Total
Number analyzed (Participants) | 1 | 0 | 1
Age Categorical [Number; unit: years]
  <=18 years | 0 |  | 0 [0 to 0]
  Between 18 and 65 years | 1 [49 to 49] |  | 1 [49 to 49]
  >=65 years | 0 |  | 0 [0 to 0]
Gender [Number; unit: participants]
  Female | 1 |  | 1
  Male | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Sleep Response of Patients
Description: Objective responses measured by wrist actigraph (measures sleep movement), and the Sp02 monitor (measures the % oxy-hemoglobin in the blood)
Time Frame: Longitudinal study with major responses measured on days 0 (day of operation) and days 1-6 post-operative
Population: Since unable to accrue an adequate number of cases with data, unable to provide analysis.
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 8 Months
Arm/Group | Melatonin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

LIMITATIONS AND CAVEATS:
Study terminated early due to low recruitment, no analysis done.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No